CLINICAL TRIAL: NCT03236480
Title: Dynamic Changes of the Respiratory Microbiota and Its Relationship to Fecal Microbiota in Chronic Obstructive Pulmonary Disease
Brief Title: The Gut-lung Axis in Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Ningde City Hospital, Fujian, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2109901; 2016YFC0903800 (Other Grant/Funding Number: Ministery of science and technology of China)
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Microbiota; Immunity, Mucosal; Metabolism
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1.Lower respiratory tract specimens including sputum, endotracheal aspiration and bronchoalveolar lavage fluid. 2.Peripheral whole blood samples 3.fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Patients who admitted to Peking Universtiy People's Hospital and Ningde City Hospital between January 2017 and January 2019 with AECOPD will be enrolled
- healthy control: People aged over 40, without any chronic respiratory disease or acute respiratory infections in the last 2 weeks, and be willing to participate in the study

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) are 2-3 times more likely to occur together with chronic gastrointestinal tract (GIT) diseases, such as inflammatory bowel disease (IBD) or irritable bowel syndrome (IBS). Similarly, despite many patients have no history of acute or chronic respiratory disease, up to 50% of IBD patients and 33% of IBS patients have pulmonary involvement, such as inflammation or impaired lung function. Increasing evidence indicated chronic gut and lung disease share key conceptual features with the disorder and dysregulation of the microbial ecosystem. However, the underlying mechanisms are not well understood.

Our study is aimed to elucidate the intimate relationship between the gastrointestinal tract and respiratory tract, and uncover the mechanisms by which the gut microbiota affects the immune responses in the lungs, and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* admitted to hospital with an exacerbation of COPD;
* with no history of probiotics taken;
* the duration of antibiotics treatment before enrollment should be less than 72 hours.

Exclusion Criteria:

* being immunocompromised, including history of glucocorticoid taken for more than 1 month, history of immunosuppressive therapy, history of human immunodeficiency virus (HIV) infection, solid tumor or hematological malignancy;
* history of long-term nursing home stays;
* history of recently hospitalized (<90 days).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Peking University People's Hospital and Ningde City Hospital with an exacerbation of COPD between January 2017 and January 2019 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | patients will be followed for 3 months after their remission from hospital
  all-cause death after the enrollment

SECONDARY OUTCOMES:
exacerbations | during the 3-month follow-up
  exacerbations of COPD

CONTACTS AND LOCATIONS:
Overall Officials: Zhancheng Gao, Pro., Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xie Y, Xue Q, Jiao W, Wu J, Yu Y, Zhao L, Xu Y, Deng X, Fang G, Zheng Y, Gao Z. Associations Between Sputum Torque Teno Virus Load and Lung Function and Disease Severity in Patients With Chronic Obstructive Pulmonary Disease. Front Med (Lausanne). 2021 Apr 22;8:618757. doi: 10.3389/fmed.2021.618757. eCollection 2021. PMID 33968949